CLINICAL TRIAL: NCT00075062
Title: Characteristics of Baseline Mucosal Indices of Injury and Inflammation in Men For Use in Rectal Microbicide Trials
Brief Title: A Study of Male Rectal Samples in Preparation for Future Rectal Microbicide Trials
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Other Study IDs: HPTN 056
Record Dates: First submitted 2003-12-31; First posted 2004-01-01 (Estimated); Last update posted 2008-08-21 (Estimated); Status verified 2006-05

CONDITIONS: HIV Infections; HIV Seronegativity
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: Flexible Sigmoidoscopy
Procedure: Rectal Biopsy

SUMMARY:
Microbicides are drugs that destroy microbes such as viruses and bacteria. Rectal microbicides may be able to prevent transmission of HIV during anal intercourse. The purpose of this study is to obtain rectal samples from men to learn information that may be valuable in future clinical trials of rectal microbicides.

DETAILED DESCRIPTION:
Rectal microbicides to prevent HIV transmission are currently being developed in the hope that someday they will be widely used to prevent sexually transmitted HIV. This study will examine variables in male rectal tissue; this information may be useful for future rectal microbicide safety and efficacy studies. The study will evaluate the differences in rectal tissue from HIV infected or uninfected males who either engage in anal-receptive sex (men who sleep with men, or MSM) or do not have anal-receptive sex.

The study will last approximately 7 months, with 6 weeks of follow-up. There are four groups in this study. Groups 1 and 2 will enroll HIV uninfected men; Groups 3 and 4 will enroll HIV infected men. Groups 1, 3, and 4 will comprise MSM who engage in anal-receptive sex; Group 2 will comprise men who do not. Patients will provide medical and medication history, undergo a complete physical exam, and receive HIV counseling at screening. An anoscopy (examination of the anus, anal canal, and lower rectum) and blood draw will be conducted at screening, study entry, and Weeks 2 and 4. Rectal secretions will be collected and a sigmoidoscopy (an internal examination of the rectum, distal sigmoid colon, and large bowel using a small camera) will be performed at study entry and Weeks 2 and 4.

ELIGIBILITY:
Inclusion Criteria for All Participants:

* HIV status confirmed by ELISA/Western Blot at screening
* CD4 count greater than 200 cells/mm3 at screening
* Able and willing to communicate in English
* Able and willing to provide adequate information for locator purposes

Inclusion Criteria for Men Practicing Anal-Receptive Sex (Groups 1, 3 and 4):

* Engaged in anal-receptive sex an average of at least once a week in the 2 months prior to study entry
* Agree to refrain from anal intercourse for 24 hours prior to and for one week after sigmoidoscopy

Inclusion Criteria for Men Not Practicing Anal-Receptive Sex (Group 2)

* No history of anal receptive intercourse in the 2 months prior to study entry

Inclusion Criteria for HIV Infected Men (Groups 3 and 4):

* Viral load of either greater than 10,000 copies of RNA/ml plasma or less than 50 copies RNA/ml plasma for at least 2 months prior to study entry
* Have not changed antiretroviral therapy within 6 weeks prior to study entry

Exclusion Criteria:

* For HIV infected patients, 3 or more HSV-2 (herpes) outbreaks in the 12 months prior to screening or 1 or more HSV-2 outbreaks in the 6 months prior to screening
* Active, serious infections (other than HIV) requiring parenteral antibiotic therapy within 15 days prior to screening
* Inflammatory bowel disease (ulcerative colitis or Crohn's disease) or rectal cancer
* Rectal surgery, including fistulectomy
* Diagnosed bleeding disorder, including hemophilia, thrombocytopenia, impaired blood clotting, or current use of anticoagulants that, in the opinion of the investigator, would make participation in the study unsafe or complicate interpretation of study outcome data
* Prosthetic heart valve or diagnosis of valve abnormality
* Hemorrhoid surgery in the 6 months prior to screening
* Bleeding hemorrhoids at screening or in the 6 weeks prior to study entry
* Anal fistulae in the 6 weeks prior to study entry
* Active diarrheal disease (greater than 3 times a day) or bleeding disorder
* Rectal cultures positive for chlamydia or gonorrhea at screening or within 1 month prior to study entry
* Unprotected anal intercourse in the 3 months prior to study entry
* Any other clinical condition or prior therapy that, in the opinion of the investigator, would make the patient unsuitable for the study or unable to comply with study requirements
* Enrolled in any other clinical trial for the duration of their participation in HPTN 056

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16

CONTACTS AND LOCATIONS:
Overall Officials: Ian McGowan, MD, PhD, Study Chair — University of California, Los Angeles; Peter Anton, MD, Study Chair — University of California, Los Angeles
Locations (1):
- David Geffen School of Medicine at UCLA, Los Angeles, California, United States

REFERENCES:
- [Background] Baron S, Poast J, Nguyen D, Cloyd MW. Practical prevention of vaginal and rectal transmission of HIV by adapting the oral defense: use of commercial lubricants. AIDS Res Hum Retroviruses. 2001 Jul 20;17(11):997-1002. doi: 10.1089/088922201300343672. PMID 11485616
- [Background] Garg S, Tambwekar KR, Vermani K, Kandarapu R, Garg A, Waller DP, Zaneveld LJ. Development pharmaceutics of microbicide formulations. Part II: formulation, evaluation, and challenges. AIDS Patient Care STDS. 2003 Aug;17(8):377-99. doi: 10.1089/108729103322277402. PMID 13678540
- [Background] Gross M, Buchbinder SP, Celum C, Heagerty P, Seage GR 3rd. Rectal microbicides for U.S. gay men. Are clinical trials needed? Are they feasible? HIVNET Vaccine Preparedness Study Protocol Team. Sex Transm Dis. 1998 Jul;25(6):296-302. doi: 10.1097/00007435-199807000-00005. PMID 9662763